CLINICAL TRIAL: NCT04295161
Title: A Study in Healthy Male Subjects Designed to Evaluate the Pharmacokinetic Profile of Abiraterone Following Administration of Immediate Release Formulations
Brief Title: A Study Designed to Evaluate the Pharmacokinetic Profile of Abiraterone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zentiva, k.s. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABIRAL00005
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Reference (Active Comparator)
  Interventions: Drug: Abiraterone Acetate
- Prototype 1 (Experimental)
  Interventions: Drug: Abiraterone Acetate
- Prototype 2 (Experimental)
  Interventions: Drug: Abiraterone Acetate
- Prototype 3 (Experimental)
  Interventions: Drug: Abiraterone Acetate
- Prototype 4 fasted (Experimental): administered in fasted state
  Interventions: Drug: Abiraterone Acetate
- Prototype 4 fed (Experimental): Administered in fed state
  Interventions: Drug: Abiraterone Acetate

INTERVENTIONS:
Drug: Abiraterone Acetate — Abiraterone acetate immediate release formulations

SUMMARY:
A Study in Healthy Male Subjects Designed to Evaluate the Pharmacokinetic Profile of Abiraterone Following Administration of Immediate Release Formulations

DETAILED DESCRIPTION:
This was a single centre, 2 part, open-label study in healthy male subjects. Parts 1 and 2 were conducted in separate cohorts of subjects; subjects were not permitted to participate in both parts. Part 1 was a part-randomised, 4 period crossover study planned to include 24 healthy male subjects. Part 2 was a randomised 2-period crossover study in 12 healthy male subjects. The aim was to evaluate the pharmacokinetic profiles of abiraterone following administration of immediate release prototype formulations in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Age 18 to 55 years of age at the time of signing informed consent
3. Expressed a desire not to father children in the near future (within 6 months of last IMP dose); males under 40 years of age must have been vasectomised
4. Body mass index (BMI) of 18.5 to 30.0 kg/m2 as measured at screening
5. Willing and able to communicate and participate in the whole study
6. Provided written informed consent
7. Agreed to adhere to the contraception requirements defined in Section 9.4 of the protocol

Exclusion Criteria:

1. Subjects who received any IMP in a clinical research study within the 3 months or 90 days prior to Day 1 Period 1
2. Males with a pregnant female partner
3. Subjects were unable or unwilling to consume the standard high-fat breakfast (Part 2)
4. Subjects were study site employees, or immediate family members of a study site or sponsor employee
5. Subjects who had previously been enrolled in this study. Subjects who had taken part in Part 1 were not permitted to take part in Part 2
6. History of any drug or alcohol abuse in the past 2 years prior to screening
7. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type) as confirmed by a repeat of the first positive alcohol breath test at screening or admission
8. Current smokers and those who had smoked within the last 12 months. A confirmed breath carbon monoxide (CO) reading of greater than 10 ppm, as confirmed by repeat of the first test at screening or admission
9. Current users of e-cigarettes and nicotine replacement products and those who had used these products within the last 12 months prior to screening
10. Subjects without suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening
11. Clinically significant abnormal biochemistry, haematology or urinalysis at screening as judged by the investigator
12. Serum potassium below the lower limit of the laboratory reference range at screening
13. Alanine aminotransferase >1.5× upper limit of laboratory reference range at screening
14. Total bilirubin >1.5× upper limit of laboratory reference range at screening
15. Confirmed positive drugs of abuse test result
16. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) orhuman immunodeficiency virus (HIV) results at screening
17. Systolic blood pressure (BP) >140 mmHg, diastolic blood pressure >90 mmHg (systolic blood pressure up to 150 mmHg allowed in subjects >45 years of age) at screening or Period 1 Day 1 pre-dose
18. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator
19. Subjects with a history of cholecystectomy or gall stones
20. Serious adverse reaction or serious hypersensitivity to any drug
21. History of any hypersensitivity reaction to abiraterone or the formulation excipients regardless of severity
22. Subjects with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption, lactose intolerance
23. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever was allowed unless it was active
24. Donation or loss of greater than 400 mL of blood within the previous 3 months prior to screening
25. Subjects who were taking, or had taken, any prescribed or over-the-counter drug (other than 4 g of paracetamol per day) or herbal remedies in the 14 days before Day 1, Period 1. Exceptions may have been applied on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI
26. Use of known strong CYP3A4 inducers, including St John's Wort, in the 30 days prior to Period 1 Day 1
27. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Abiraterone Cmax | 24h
  maximal concentration of abiraterone in human plasma
Abiraterone AUC | 24h
  total exposure up to 24h of abiraterone in human plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: No